CLINICAL TRIAL: NCT01924156
Title: Safety and Therapeutic Efficacy of DC Vaccine Combined With Cytokine-induced Killer Cells in Patients With Renal Cell Carcinoma: a Phase I/II Study
Brief Title: DC Vaccine Combined With CIK Cells in Patients With Renal Cell Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-CTC-DC/CIK-RCC
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adenovirus-transfected DC + CIK (Experimental): adenovirus-transfected autologous DC vaccine plus CIK cells
  Interventions: Biological: adenovirus-transfected DC + CIK

INTERVENTIONS:
Biological: adenovirus-transfected DC + CIK — adenovirus-transfected DC vaccine plus CIK cells

SUMMARY:
The aim of this Phase I/II study is to evaluate the safety and efficacy of dendritic cells (DC) vaccine combined with cytokine-induced killer (CIK) cells in patients with renal cell carcinoma. Experimental recombinant adenovirus-transfected DC, which engineered to express MUC1 and Survivin are used for DC-based immunotherapy. Based on the results of our previously performed preclinical study with DC vaccine combined with CIK cells, the investigators plan to perform the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years at time of consent
* Histopathologically confirmed diagnosis of renal cell carcinoma
* Received standardized treatment of renal cell carcinoma
* Interval between the last standardized treatment and DC/CIK treatment ≥ 4weeks
* KPS (Karnofsky performance scale) >60
* Patient's written informed consent
* Predicted survival >3 months
* No severe viral or bacterial infections

Exclusion Criteria:

* Receiving chemotherapy, radiotherapy or other therapy
* Patients with other malignancies and infectious diseases
* Pregnant and breast-feeding patient
* Currently participating in another clinical trial
* Unfit for participating in this clinical trial in investigators' opinions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
objective tumor response (CR+PR) as measured by RECIST criteria | 4 weeks after DC/CIK treatment

SECONDARY OUTCOMES:
number of participants with adverse events | 3 days within DC/CIK treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hu Chen, M.D., Ph.D., Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Department of Hematopoietic Stem Cell Transplantation, Beijing, China

REFERENCES:
- [Derived] Wang D, Zhang B, Gao H, Ding G, Wu Q, Zhang J, Liao L, Chen H. Clinical research of genetically modified dendritic cells in combination with cytokine-induced killer cell treatment in advanced renal cancer. BMC Cancer. 2014 Apr 10;14:251. doi: 10.1186/1471-2407-14-251. PMID 24720900